CLINICAL TRIAL: NCT04209972
Title: The Benefit of Ultra-high Resolution Computed Tomography: Precision of Repeated Volume Measurements of Pulmonary Nodules
Brief Title: The Benefit of UHR-CT: Precision of Repeated Volume Measurements of Pulmonary Nodules
Acronym: Coffee Break
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL67905.091.18
Record Dates: First submitted 2019-03-20; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Nodule, Solitary
Keywords: Ultra-high resolution CT; volume measumerents
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Intervention Model Description: 2 groups, 40 patients on one CT scanner, 40 different patients on the other CT scanner.
Who Masked: Participant
Masking Description: Patients does not know if he is on the standard CT scanner, or on the UHR CT scanner
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients on CT1 (Active Comparator): Patients will undergo two pre-contrast scans, and will be in between the two scans be off and on the table at a standard CT scanner. (Aquilion One Genesis, Canon Medical Systems)
  Interventions: Device: Genesis high-end CT scanner
- Patients on CT2 (Active Comparator): Patients will undergo two pre-contrast scans, and will be in between the two scans be off and on the table at a UHRCT scanner. (Aquilion One Precision, Canon Medical Systems)
  Interventions: Device: Precision Ultra-High-Resolution CT scanner

INTERVENTIONS:
Device: Precision Ultra-High-Resolution CT scanner — Patients will be divided on one of the two CT scanners. This group will be scanned on the Precision CT scanner.
  Arms: Patients on CT2
Device: Genesis high-end CT scanner — Patients will be divided on one of the two CT scanners. This group will be scanned on the Aquilion one Genesis.
  Arms: Patients on CT1

SUMMARY:
To assess the variability of semi-automated volume measurements of pulmonary nodules on same-day repeated scans of equal radiation dose from two different CT scanners: One high-end CT scanner with standard spatial resolution (CT1) and one UHRCT scanner (CT2), in patients with known or suspected pulmonary metastases.

DETAILED DESCRIPTION:
Rationale: Ultra-high resolution computed tomography (UHRCT) produces radiological images with a spatial resolution of 0.25 mm in a matrix of 1024x1024. This should decrease measurement variation of nodule growth as a marker of malignancy, by making nodule delineation more precise for automatic volumetry segmentation and volume doubling time assessment than in conventional CT. If possible, this can shorten follow up of incidental pulmonary nodules to exclude malignancy, with less medicalisation and patient anxiety.

Objective: To assess the variability of semi-automated volume measurements of pulmonary nodules in patients with known or suspected pulmonary metastases on same-day repeated scans of equal radiation dose from two different CT scanners: CT scanner with standard spatial resolution (conventional CT, CT1) and UHRCT (CT2).

Study design: This is a single center prospective trial on 80 patients with known or suspected pulmonary metastases who are scheduled for chest and/or abdominal CT. Study participants will undergo two additional partial chest CT scans on either CT 1 or CT 2 for research purpose only, at similar radiation dose. Patients are equally divided across CT 1 and 2.

Study population: Patients who are 18 years or older with known solid pulmonary nodules compatible with metastases and who are willing and able to give informed consent are eligible. Patients are excluded if they have less than two eligible pulmonary nodules with a z range of 16 cm. Nodules with calcifications, surrounding opacities, or vessel- or pleural abutment will be excluded from analysis.

Main study parameters/endpoints: The main endpoint of this study is the upper limit of the 95% confidence interval of repeated semi-automated nodule volume measurements of both CT scanners.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

CT imaging is associated with risks related to the use of ionizing radiation. The CT protocol including the scheduled CT scan and the additional scans in this study has been carefully designed to have a total radiation dose at the same level as the achievable diagnostic reference level of chest CT in the Netherlands, which is 542 mGycm in 2013 (1). The burden associated with the two extra study CT acquisitions comprises a dose length product (DLP) of 120.4 mGy•cm for research (1.7 mSv, which is lower than the background radiation of one year in the Netherlands, with a conversion factor of 0.014 from Deak et al (2)).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* A solid primary tumour anywhere in the body and solid, noncalcified nodules in the pulmonary parenchyma on previous CT scans suspected for pulmonary metastases, according to radiological reports
* Two lung nodules that do not abut vessels or pleura with a two dimensional diameter between 5 and 10 mm within a distance of each other of 16 cm in the craniocaudal direction

Exclusion Criteria:

* Immobility (not able to stand up and get off the scanner table)
* Patients who received local pulmonary treatment: Radiotherapy, Excision, Ablation
* Patients with radiologically suspected lymphangitis carcinomatosa or consolidations around the nodules.
* Patients who only have calcified pulmonary nodules or nodules that abut vessels or pleura.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
The main endpoint of this study is the difference in precision in millimeter between the two CT scanners. | 4 months
  The precision of each scanner is obtained by the standard deviation between the two measurements. The difference between scanners is tested with an F-test and the precision of each scanner is shown by a Bland-Altman plot

SECONDARY OUTCOMES:
Evaluation of image quality (segmentation errors) | 5 months
  Evaluate the image quality of the scans
Evaluation of image quality (motion artefacts) | 5 months
  Evaluate the image quality of the scans

OTHER OUTCOMES:
Patient characteristics (age) | 4 months
  Patient characteristics (age)
Patient characteristics (height) | 4 months
  Patient characteristics (height)
Patient characteristics (weight) | 4 months
  Patient characteristics (weight)
Radiation dose | 4 months
  Radiation dose

CONTACTS AND LOCATIONS:
Overall Officials: Monique Brink, PhD, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet

REFERENCES:
- [Result] van der Molen AJ, Schilham A, Stoop P, Prokop M, Geleijns J. A national survey on radiation dose in CT in The Netherlands. Insights Imaging. 2013 Jun;4(3):383-90. doi: 10.1007/s13244-013-0253-9. Epub 2013 May 15. PMID 23673455
- [Result] Deak PD, Smal Y, Kalender WA. Multisection CT protocols: sex- and age-specific conversion factors used to determine effective dose from dose-length product. Radiology. 2010 Oct;257(1):158-66. doi: 10.1148/radiol.10100047. PMID 20851940
- [Result] Alpert JB, Ko JP. Management of Incidental Lung Nodules: Current Strategy and Rationale. Radiol Clin North Am. 2018 May;56(3):339-351. doi: 10.1016/j.rcl.2018.01.002. Epub 2018 Mar 7. PMID 29622070
- [Result] MacMahon H, Naidich DP, Goo JM, Lee KS, Leung ANC, Mayo JR, Mehta AC, Ohno Y, Powell CA, Prokop M, Rubin GD, Schaefer-Prokop CM, Travis WD, Van Schil PE, Bankier AA. Guidelines for Management of Incidental Pulmonary Nodules Detected on CT Images: From the Fleischner Society 2017. Radiology. 2017 Jul;284(1):228-243. doi: 10.1148/radiol.2017161659. Epub 2017 Feb 23. PMID 28240562
- [Result] Baldwin DR, Callister ME; Guideline Development Group. The British Thoracic Society guidelines on the investigation and management of pulmonary nodules. Thorax. 2015 Aug;70(8):794-8. doi: 10.1136/thoraxjnl-2015-207221. Epub 2015 Jul 1. PMID 26135833
- [Result] Devaraj A, van Ginneken B, Nair A, Baldwin D. Use of Volumetry for Lung Nodule Management: Theory and Practice. Radiology. 2017 Sep;284(3):630-644. doi: 10.1148/radiol.2017151022. PMID 28825886
- [Result] Wormanns D, Kohl G, Klotz E, Marheine A, Beyer F, Heindel W, Diederich S. Volumetric measurements of pulmonary nodules at multi-row detector CT: in vivo reproducibility. Eur Radiol. 2004 Jan;14(1):86-92. doi: 10.1007/s00330-003-2132-0. Epub 2003 Nov 13. PMID 14615902
- [Result] Gietema HA, Schaefer-Prokop CM, Mali WP, Groenewegen G, Prokop M. Pulmonary nodules: Interscan variability of semiautomated volume measurements with multisection CT-- influence of inspiration level, nodule size, and segmentation performance. Radiology. 2007 Dec;245(3):888-94. doi: 10.1148/radiol.2452061054. Epub 2007 Oct 8. PMID 17923508
- [Result] Goodman LR, Gulsun M, Washington L, Nagy PG, Piacsek KL. Inherent variability of CT lung nodule measurements in vivo using semiautomated volumetric measurements. AJR Am J Roentgenol. 2006 Apr;186(4):989-94. doi: 10.2214/AJR.04.1821. PMID 16554568
- [Result] Hein PA, Romano VC, Rogalla P, Klessen C, Lembcke A, Bornemann L, Dicken V, Hamm B, Bauknecht HC. Variability of semiautomated lung nodule volumetry on ultralow-dose CT: comparison with nodule volumetry on standard-dose CT. J Digit Imaging. 2010 Feb;23(1):8-17. doi: 10.1007/s10278-008-9157-5. Epub 2008 Sep 5. PMID 18773240
- [Result] Han D, Heuvelmans MA, Oudkerk M. Volume versus diameter assessment of small pulmonary nodules in CT lung cancer screening. Transl Lung Cancer Res. 2017 Feb;6(1):52-61. doi: 10.21037/tlcr.2017.01.05. PMID 28331824
- [Result] Tanaka R, Yoshioka K, Takagi H, Schuijf JD, Arakita K. Novel developments in non-invasive imaging of peripheral arterial disease with CT: experience with state-of-the-art, ultra-high-resolution CT and subtraction imaging. Clin Radiol. 2019 Jan;74(1):51-58. doi: 10.1016/j.crad.2018.03.002. Epub 2018 Apr 5. PMID 29627067
- [Result] Zhou W, Montoya J, Gutjahr R, Ferrero A, Halaweish A, Kappler S, McCollough C, Leng S. Lung Nodule Volume Quantification and Shape Differentiation with an Ultra-High Resolution Technique on a Photon Counting Detector CT System. Proc SPIE Int Soc Opt Eng. 2017 Feb 11;10132:101323Q. doi: 10.1117/12.2255736. Epub 2017 Mar 9. PMID 28392613
- [Result] de Hoop B, Gietema H, van Ginneken B, Zanen P, Groenewegen G, Prokop M. A comparison of six software packages for evaluation of solid lung nodules using semi-automated volumetry: what is the minimum increase in size to detect growth in repeated CT examinations. Eur Radiol. 2009 Apr;19(4):800-8. doi: 10.1007/s00330-008-1229-x. Epub 2008 Nov 19. PMID 19018537
- [Result] Leng S, Gutjahr R, Ferrero A, Kappler S, Henning A, Halaweish A, Zhou W, Montoya J, McCollough C. Ultra-High Spatial Resolution, Multi-Energy CT using Photon Counting Detector Technology. Proc SPIE Int Soc Opt Eng. 2017 Feb 11;10132:101320Y. doi: 10.1117/12.2255589. Epub 2017 Mar 9. PMID 28392615
- [Result] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Result] Kalra MK, Sodickson AD, Mayo-Smith WW. CT Radiation: Key Concepts for Gentle and Wise Use. Radiographics. 2015 Oct;35(6):1706-21. doi: 10.1148/rg.2015150118. PMID 26466180